CLINICAL TRIAL: NCT02093637
Title: Rapid Extremity Pain Relief by Battlefield Acupuncture After Orthopedic Surgery: A Randomized Clinical Trial
Brief Title: Rapid Extremity Pain Relief by Battlefield Acupuncture After Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDG20120024H
Record Dates: First submitted 2013-07-11; First posted 2014-03-21 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo acupuncture (Placebo Comparator): Placebo acupuncture up to 5 acupuncture needles* in each ear (up to 10 needles total) at points identified by point-finder to have no electrical conductance) plus usual operative and post-operative care (narcotic and non-narcotic pain medication).
  Interventions: Other: Placebo acupuncture
- Battlefield Acupuncture (Experimental): Usual operative and post-operative care (narcotic and non-narcotic pain medication) plus Battlefield Acupuncture (up to 5 acupuncture needles* in each ear (up to 10 needles total), identified by a point-finder.
  Interventions: Other: Battlefield Acupuncture
- standard therapy (No Intervention): standard therapy

INTERVENTIONS:
Other: Placebo acupuncture — Placebo Comparator
  Other Names: ASP needles
  Arms: Placebo acupuncture
Other: Battlefield Acupuncture — Experimental
  Other Names: ASP needles
  Arms: Battlefield Acupuncture

SUMMARY:
The purpose of this study is to determine if the addition of Battlefield Auricular Acupuncture (BFA) to standard therapy causes reduction in pain, medication use, time to ambulation without assistance, hours missed from work and increases quality of life after lower extremity surgery at two Air Force Medical Centers.

DETAILED DESCRIPTION:
We will recruit 429subjects into this research study, for an expected 309 completing the study. We estimate 120 subjects will either withdraw consent or become ineligible for the study. Subjects will be ≥18 years or older and scheduled for lower extremity surgery. To randomize subjects, we will employ a random number generator, which will minimize difference between study groups. Additionally, we will collect data about patients' length of hospital stay, which will allow for statistical control of the variable, complexity of surgical procedure. The Research Assistants/Coordinators will be responsible for obtaining Informed Consent and HIPAA Authorization from subjects, collecting data, and de-identifying data prior to review and analysis by the Investigators. The Investigators will be responsible for ongoing protocol monitoring, insertion of needles, verifying inclusion/exclusion criteria, and analyzing data.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion Criteria:

Male and female subjects (DoD beneficiaries), 18 years or older who are scheduled for lower extremity surgery below the hip.

Exclusion Criteria:

Pregnant or breastfeeding Absence of their ear Active cellulitis of their ear Ear anatomy precluding identification of acupuncture landmarks Non-English speaking Use of Hearing Aids that preclude the insertion of ASP needles Inability to comply with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Pain score | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, MD, Principal Investigator — MOFMC
Locations (2):
- United States (2):
  - David Grant Medical Center, Travis Air Force Base, California
  - Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada